CLINICAL TRIAL: NCT05803421
Title: A Phase 3, Open-Label Study of Once Daily LY3502970 Compared With Insulin Glargine in Adult Participants With Type 2 Diabetes and Obesity or Overweight at Increased Cardiovascular Risk
Brief Title: A Study of Daily Oral Orforglipron (LY3502970) Compared With Insulin Glargine in Participants With Type 2 Diabetes and Obesity or Overweight at Increased Cardiovascular Risk
Acronym: ACHIEVE-4
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18563; J2A-MC-GZGS (Other: Eli Lilly and Company); 2022-502833-25-00 (Other: EU Trial Number); U1111-1285-6821 (Other: Universal Trial Number (UTN))
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; Obesity; Overweight or Obesity; Overweight; Cardiovascular Diseases; Chronic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight; Cardiovascular Diseases; Renal Insufficiency, Chronic | interventions — orforglipron; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orforglipron (Experimental): Participants will receive escalated doses of orforglipron orally.
  Interventions: Drug: Orforglipron
- Insulin Glargine (Active Comparator): Participants will receive insulin glargine subcutaneously (SC). Doses will be individualized and titrated according to a treat-to-target algorithm.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Orforglipron — Administered orally once daily
  Other Names: LY3502970
  Arms: Orforglipron
Drug: Insulin Glargine — Administered SC once daily
  Arms: Insulin Glargine

SUMMARY:
The main purpose of this study is to determine safety and efficacy of orforglipron compared with insulin glargine in participants with type 2 diabetes and obesity or overweight at increased cardiovascular risk. The study will last approximately 2 years may include up to 27 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with type 2 diabetes mellitus (T2DM)
* Are at least 18 years of age or legal age of consent in the jurisdiction in which the study is taking place, whichever is older.
* Have HbA1c at screening

  * ≥7.0% and ≤10.5% if background diabetes medication does not include a sulfonylurea, or
  * ≥7.5% and ≤10.5% if background diabetes medication includes a sulfonylurea.
* Are on stable treatment of at least 1 and no more than 3 oral antihyperglycemic drugs for at least 90 days before screening. Antihyperglycemic drugs may include metformin, SGLT-2 inhibitors, and/or sulfonylureas
* Have increased risk for cardiovascular (CV) events due to:

  * Coronary heart disease
  * Peripheral arterial disease, presumed to be of atherosclerotic origin
  * Cerebrovascular disease, presumed to be of atherosclerotic origin
  * Chronic kidney disease (CKD)
  * Congestive heart failure (CHF) New York Heart Association (NYHA) functional classification II to III
* Are of stable weight (± 5%) for at least 90 days prior to screening
* Have a BMI ≥25 kilograms per meter squared (kg/m2) at screening

Exclusion Criteria:

* Have type 1 diabetes mellitus
* Have had chronic or acute pancreatitis any time prior to screening
* Currently receiving or planning to receive treatment for diabetic retinopathy and/or macular edema (e.g. laster photocoagulation or intravitreal injections of anty-VEGF inhibitors
* Have a known clinically significant gastric emptying abnormality
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease, or blood alanine transaminase (ALT) or aspartate aminotransferase (AST) enzyme level ≥5.0 times the upper limit of normal (ULN) for the reference range, as determined by the central laboratory
* Have had any of the following within 60 days prior to screening: acute myocardial infarction, cerebrovascular accident (stroke), or hospitalization for congestive heart failure
* Have an eGFR <15 mL/min/1.73 m2 as determined at screening
* Have a family (first-degree relative) or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
* Have been taking any other diabetes medicines other than metformin, SGLT-2 inhibitors, and/or sulfonylureas during the last 90 days
* Have used any weight loss drugs, including herbal or nutritional supplements, within 90 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2749 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of Any Major Adverse Cardiovascular Event (MACE-4) [Myocardial Infarction (MI), Stroke, Hospitalization for Unstable Angina, or Cardiovascular (CV) Death] | Baseline to End of the Study (Approximate Maximum 104 Weeks)
  Time to First Occurrence of Any MACE-4 (Myocardial Infarction (MI), Stroke, Hospitalization for Unstable Angina, or Cardiovascular [CV] Death)

SECONDARY OUTCOMES:
Time to First Occurrence of Any MACE-3 Event (MI, Stroke, or CV death) | Baseline to End of the Study (Approximately 104 Weeks)
  Time to First Occurrence of Any MACE-3 Event (MI, Stroke, or CV death)
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 52
  Change from Baseline in HbA1c
Change from Baseline in Fasting Serum Glucose | Baseline, Week 52
  Change from Baseline in Fasting Serum Glucose
Change from Baseline in Daily Average 7-point Self-monitoring Blood Glucose (SMBG) Profile | Baseline, Week 52
  Change from Baseline in Daily Average 7-point SMBG
Percentage of Participants with HbA1c Target Values Less Than (<)7.0% (53 mmol/mol) | Week 52
  Percentage of Participants with HbA1c Target Values <7.0% (53 mmol/mol)
Change from Baseline in Body Weight | Baseline, Week 52
  Change from Baseline in Body Weight
Percent Change from Baseline Body Weight | Week 52
  Percent Change from Baseline Body Weight
Change from Baseline in Short Form 36 Version 2 (SF-36v2) Acute Form Domain Score | Baseline, Week 52
  The SF-36v2 acute form is a 36-item generic, participant completed measure designed to assess 8 domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Scores of each domain are measured by T-scores, with a mean of 50 and standard deviation of 10; higher scores indicate better levels of function and/or better health.
Pharmacokinetics (PK): Plasma Serum Concentrations of Orforglipron | Baseline through Week 52
  PK will be estimated based on the population PK model.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (358):
- United States (173):
  - Alliance for Multispecialty Research, LLC, Daphne, Alabama
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - Cahaba Research - Pelham, Pelham, Alabama
  - Syed Research Consultants Llc, Sheffield, Alabama
  - The Institute for Liver Health, Chandler, Arizona
  - Aventiv Research, Mesa, Arizona
  - Arizona Liver Health - Peoria, Peoria, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Absolute Clinical Research, Phoenix, Arizona
  - Clinical Research Institute of Arizona (CRI) - Sun City West, Sun City West, Arizona
  - Alliance for Multispecialty Research, LLC, Tempe, Arizona
  - Orange Grove Family Practice, Tucson, Arizona
  - KLR Business Group, Inc. dba Arkansas Clinical Research, Little Rock, Arkansas
  - Hope Clinical Research, Inc., Canoga Park, California
  - Valley Clinical Trials, Inc., Covina, California
  - Neighborhood Healthcare Institute of Health, Escondido, California
  - Valley Research, Fresno, California
  - Orange County Research Center, Lake Forest, California
  - Ark Clinical Research, Long Beach, California
  - Pacific Clinical Studies, Los Alamitos, California
  - Velocity Clinical Research, Los Angeles, Los Angeles, California
  - Infinity Clinical Research - Norco, Norco, California
  - Velocity Clinical Research, North Hollywood, North Hollywood, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Rancho Cucamonga Clinical Research, Rancho Cucamonga, California
  - LCGK Research, San Carlos, California
  - Norcal Endocrinology & Internal Medicine, San Ramon, California
  - Velocity Clinical Research, Coastal Heart Medical Group, Santa Ana, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Millennium Clinical Trials, Westlake Village, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Legacy Clinical Trials, Colorado Springs, Colorado
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Orlando Heart & Vascular Institute, Altamonte Springs, Florida
  - JEM Research Institute, Atlantis, Florida
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Velocity Clinical Research, New Smyrna Beach, Edgewater, Florida
  - Alliance for Multispecialty Research, LLC, Fort Myers, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Nature Coast Clinical Research - Inverness, Inverness, Florida
  - Northeast Research Institute - Downtown Office, Jacksonville, Florida
  - Clinical Research of Central Florida, Lakeland, Florida
  - Clinical Site Partners Leesburg, Leesburg, Florida
  - L&C Professional Medical Research Institute, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Adult Medicine of Lake County, Mt. Dora, Florida
  - Renstar Medical Research, Ocala, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Better Life Clinical Research, Tampa, Florida
  - Precision Research Center, Tampa, Florida
  - Care Access - Tampa, Tampa, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Encore Medical Research - Weston, Weston, Florida
  - Conquest Research, Winter Park, Florida
  - Balanced Life Health Care Solutions/SKYCRNG, Lawrenceville, Georgia
  - The Jones Center Clinical Research, Macon, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - Saltzer Health, Nampa, Idaho
  - Elite Clinical Trials, Rexburg, Idaho
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Midwest CRC, Crystal Lake, Illinois
  - AMR Clinical, Oak Brook, Illinois
  - NorthShore University Health System, Skokie, Illinois
  - American Health Network of Indiana, LLC - Avon, Avon, Indiana
  - Investigators Research Group, Brownsburg, Indiana
  - Qualmedica Research, LLC, Evansville, Indiana
  - American Health Network of Indiana, LLC - Franklin, Franklin, Indiana
  - American Health Network of Indiana, LLC - Greenfield, Greenfield, Indiana
  - American Health Network of Indiana, LLC - Muncie, Muncie, Indiana
  - University of Iowa, Iowa City, Iowa
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - Cotton O'Neil Mulvane, Topeka, Kansas
  - Qualmedica Research, Bowling Green, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Louisiana Heart Center - Convington, Covington, Louisiana
  - Care Access - Lake Charles (Bayou Pines), Lake Charles, Louisiana
  - Alliance for Multispecialty Research, LLC, New Orleans, Louisiana
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Revival Research Institute, Dearborn, Michigan
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - SKY Clinical Research Network Group - Hall, Fayette, Mississippi
  - SKY Integrative Medical Center/SKYCRNG, Ridgeland, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - Diabetes and Endocrinology Specialists, Chesterfield, Missouri
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Logan Health Research, Kalispell, Montana
  - Montana Medical Research, Missoula, Montana
  - Sierra Clinical Research, Las Vegas, Nevada
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Palm Research Center Sunset, Las Vegas, Nevada
  - Northern Nevada Endocrinology, Reno, Nevada
  - Renown South Meadows Medical Center, Reno, Nevada
  - UniMed Center, East Brunswick, New Jersey
  - IMA Clinical Research, Albuquerque, New Mexico
  - Albany Stratton VA Medical Center, Albany, New York
  - Meridian Clinical Research, LLC, Binghamton, New York
  - SUNY Downstate Health Sciences University, Brooklyn, New York
  - Velocity Clinical Research, Syracuse, East Syracuse, New York
  - IMA Clinical Research Westchester, Hartsdale, New York
  - NYC Research INC, Long Island City, New York
  - Mid Hudson Medical Research, New Windsor, New York
  - IMA Clinical Research Manhattan, New York, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Care Access - Fayetteville, Fayetteville, North Carolina
  - PharmQuest Life Sciences, LLC, Greensboro, North Carolina
  - Lucas Research, Inc, Morehead City, North Carolina
  - Carolina Research Center, Shelby, North Carolina
  - Accellacare - Piedmont, Statesville, North Carolina
  - Accellacare - Wilmington - 1917 Tradd Court, Wilmington, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Remington-Davis, Inc, Columbus, Ohio
  - Tekton Research, Inc, Moore, Oklahoma
  - Central States Research, Tulsa, Oklahoma
  - Northwest Research Center, Portland, Oregon
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Capital Area Research - Newport, Newport, Pennsylvania
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Preferred Clinical Research-St. Clair, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - The Research Center of The Upstate, Greenville, South Carolina
  - Care Access - Mauldin, Mauldin, South Carolina
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - New Phase Research and Development, Knoxville, Tennessee
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - South Texas Clinical Research, Corpus Christi, Texas
  - Thyroid, Endocrinology, and Diabetes, Dallas, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Cardio Voyage, Denison, Texas
  - Soma Clinical Trials, Denison, Texas
  - Care United Research, Forney, Texas
  - Diabetes and Thyroid Center of Ft. Worth, Fort Worth, Texas
  - Valley Institute of Research - Fort Worth, Fort Worth, Texas
  - Victorium Clinical Research - Houston, Houston, Texas
  - Juno Research, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Endocrine Ips, Pllc, Houston, Texas
  - Research Physicians Network, LLC, Houston, Texas
  - Biopharma Informatic, LLC, McAllen, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Texas Diabetes & Endocrinology, P.A., Round Rock, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Soma Clinical Trials, Wylie, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Chrysalis Clinical Research, St. George, Utah
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Kalo Clinical Research, West Valley City, Utah
  - Manassas Clinical Research Center, Manassas, Virginia
  - Virginia Research Center, Midlothian, Virginia
  - Eastern Virginia Medical School (EVMS) Strelitz Diabetes Research Center, Norfolk, Virginia
  - Centricity Research Suffolk Family Medicine, Suffolk, Virginia
  - Eastside Research Associates, Redmond, Washington
  - MultiCare Rockwood Clinic- Main, Spokane, Washington
  - Universal Research Group, Tacoma, Washington
  - St. Vincent Hospital d/b/a Prevea Health, Green Bay, Wisconsin
  - Clinical Investigation Specialists, Kenosha, Wisconsin
- Argentina (16):
  - Buenos Aires Macula S.A, Buenos Aires
  - CEMEDIC, Buenos Aires
  - Centro Privado de Medicina Familiar / Mindout Research, Buenos Aires
  - Cardiología Palermo, Buenos Aires
  - CIPREC, Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Glenny Corp. S.A., Buenos Aires
  - CENUDIAB, Buenos Aires
  - Organizacion Medica de Investigacion, CABA
  - Hospital San Roque, Córdoba
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - Polo de Salud Vistalba, Luján de Cuyo
  - Instituto Médico Catamarca IMEC, Rosario
  - Investigaciones Clínicas Tucumán, San Miguel de Tucumán
- Austria (9):
  - Krankenhaus St. Josef Braunau, Braunau am Inn
  - VIVIT, Feldkirch
  - Medizinische Universität Graz, Graz
  - Konventhospital der Barmherzigen Brüder Linz, Linz
  - Private Practice - Dr. Evelyn Fliesser-Gorzer, Sankt Stefan ob Stainz
  - Klinik Landstraße, Vienna
  - Zentrum für klinische Studien Dr Hanusch Gmbh, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Klinik Hietzing, Vienna
- Brazil (18):
  - Centro de Pesquisa Clinica do Coracao, Acaraju
  - Centro de Pesquisa Clinica do Brasil, Brasília
  - Hospital Brasilia, Brasília
  - Instituto de Pesquisa clinica de Campinas, Campinas
  - Centro de Pesquisa Sao Lucas, Campinas
  - Loema Instituto de Pesquisa Clinica, Campinas
  - Instituto de Estudos e Pesquisas Clinicas do Ceara IEP-CE, Fortaleza
  - Hospital Moinhos de Vento, Porto Alegre
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - Pesquisare Saude, Santo André
  - ISPEM - Instituto São José dos Campos em Pesquisas Médicas, São José dos Campos
  - CPCLIN, São Paulo
  - NotreDame Intermedica Saude S.A, São Paulo
  - BR Trials - Ensaios Clinicos e Consultoria, São Paulo
  - Hospital 9 De Julho, São Paulo
  - Instituto Dante Pazzanese de Cardiology, São Paulo
  - CEDOES, Vitória
- Czechia (21):
  - Diacentrum Brandys n.L. s.r.o., Brandýs nad Labem
  - EFERTUS healthcare s.r.o., Brno-Židenice
  - EDUMED - Broumov, Broumov
  - Nemocnice Cesky Krumlov, Český Krumlov
  - AIDIN VK s.r.o., Hranice
  - EDUMED - Jaroměř, Jaroměř
  - MUDr. Tomas Edelsberger, Krnov
  - EDUMED - Náchod, Náchod
  - PreventaMed, Olomouc
  - Private Practice - Dr. Miroslav Koliba, Ostrava
  - Diahelp s.r.o, Pardubice V
  - Dialine - Interni a diabetologicka ambulance, Pilsen
  - DiaVize s.r.o., Prague
  - MEDICON, Prague
  - MUDr. Michala Pelikanova s.r.o., Prague
  - Milan Kvapil s.r.o., Diabetologicka ambulance, Prague
  - EUC Klinika Praha, Prague
  - Praglandia s.r.o, Prague
  - FLEDIP s.r.o., Prague
  - Nefromed, Prague
  - MUDr. Barbora Diepoltova, Praha 9 - Klanovice
- Germany (11):
  - Diabetespraxis Dr. Braun, Berlin
  - Gemeinschaftspraxis für Diabetologie, Eisenach
  - Praxis am Markt - Dr. Bernd Becker, Essen
  - MVZ im Altstadt-Carree Fulda GmbH, Fulda
  - Schwerpunktpraxis für Diabetes Hormone & Stoffwechsel, Hof
  - Gemeinschaftspraxis Dr. Taeschner/Dr. Bonigut, Leipzig
  - SMO.MD GmbH, Magdeburg
  - Gemeinschaftpraxis Dr. med. Martin Prohaska und Dr. med. Felix Schulte, Mühldorf
  - RED-Institut GmbH, Oldenburg
  - Diabetologische Schwerpunktpraxis Marck Linn Pickel, Pohlheim
  - Praxis Dr. Veronika Wenzl-Bauer, Rehlingen
- Greece (6):
  - General Hospital of Athens "G. Gennimatas", Athens
  - General Hospital of Athens Laiko, Athens
  - Attikon General University Hospital, Chaïdári
  - General Hospital of Lamia, Lamia
  - Iatriko Paleou Falirou Medical Center, Palaió Fáliro
  - G. Gennimatas General Hospital of Thessaloniki, Thessaloniki
- India (11):
  - V.S. General Hospital, Ahmedabad
  - Victoria Hospital, Bangalore Medical College And Research Institute, Bangalore
  - Life Care Hospital and Research Centre, Bangalore
  - S C B Medical College and Hospital, Cuttack
  - Apollo Excelcare Hospital, Guwahati
  - Karnataka Institute of Medical Sciences, Hubli
  - Eternal Heart Care Center and Research Institute, Jaipur
  - King Edward Memorial Hospital & Seth Gordhandas Sunderdas Medical College, Mumbai
  - Central India Cardiology and Research Institute, Nagpur
  - Chellaram Diabetes Institute, Pune
  - Nirmal Hospital Pvt Ltd., Surat
- Italy (10):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - AOU Renato Dulbecco, Catanzaro
  - Università degli Studi Gabriele D' Annunzio, Chieti
  - Ospedale San Raffaele, Milan
  - University of Naples Federico II, Naples
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara
  - AO Santa Maria della Misericordia, Perugia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliero Universitaria Senese, Siena
  - Azienda sanitaria universitaria giuliano isontina ASUGI Ospedale Maggiore- Università di Trieste, Trieste
- Mexico (12):
  - Clínica San Cosme, Aguascalientes
  - Centro de Investigación Cardiometabólica de Aguascalientes, Aguascalientes
  - Investigacion En Salud Y Metabolismo Sc, Chihuahua City
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Ciudad Madero
  - Centro Para El Desarrollo de La Medicina Y de Asistencia Medica Especializada S.C., Culiacán
  - Lahoja. Asociacion Para La Investigacion Y La Farmacovigilancia, Durango
  - Diseno y Planeacion en Investigacion Medica, Guadalajara
  - Private Practice - Dr. Francisco Gerardo Padilla, Guadalajara
  - Instituto Cardiovascular de León S.C., León
  - Cardiolink Clin Trials, Monterrey
  - Centro de Estudios Clínicos de Querétaro (CECLIQ), Querétaro
  - Centro de Investigacion Cardiovascular y Metabólica, Tijuana
- Puerto Rico (9):
  - Centro de Endocrinologia y Nutricion, Caguas
  - Dorado Medical Complex, Dorado
  - Manati Center for Clinical Research, Manatí
  - Puerto Rico Medical Research, Ponce
  - Research and Cardiovascular Corp., Ponce
  - GCM Medical Group, PSC - Hato Rey Site, San Juan
  - Mindful Medical Research, San Juan
  - Mgcendo Llc, San Juan
  - Wellness clinical Research Vega Baja, Vega Baja
- Romania (19):
  - CMI Dr.Pletea Noemi SRL, Bacau
  - SC Minimed SRL, Bacau
  - Mariodiab Clinic, Brasov
  - C.M.D.T.A. Neomed, Brasov
  - Nicodiab, Bucharest
  - Geea Medical Easy Diet, Bucharest
  - Hightech Medical Services SRL-Centrul pentru Studiul Metabolismului, Bucharest
  - Centrul Medical NutriLife, Bucharest
  - Centrul Medical Endocrinologie si Diabet Dr. Paveliu, Bucharest
  - Milena Sante, Galați
  - Diamed Obesity, Galați
  - Centrul Medical Consultmed, Iași
  - Cardiomed Iași, Iași
  - Diabdana, Oradea
  - Centrul Medical Grandmed, Oradea
  - Diabmed Dr. Popescu Alexandrina, Ploieşti
  - Clinica Korall, Satu Mare
  - Centrul Medical Mediab, Târgu Mureş
  - Cabinet Medical Dr.Geru, Timișoara
- Slovakia (11):
  - Diacrin s.r.o., Bratislava
  - Diab - Int, Bytča
  - Human Care s.r.o., Košice
  - IN-DIA, Lučenec
  - NEDÚ - Národný endokrinologický a diabetologický ústav n.o., Ľubochňa
  - MediVet s.r.o., Malacky
  - DIA-MED CENTRUM s.r.o., Púchov
  - Tatratrial s.r.o., Rožňava
  - MEDI-DIA s.r.o., Sabinov
  - Areteus s.r.o., Trebišov
  - JAL, Trnava
- South Korea (13):
  - Eulji University Hospital, Daejeon
  - Hanyang University Guri Hospital, Guri-si
  - Yeungnam Univeristy Medical Center, Gyeongsan-si
  - Seoul National University Bundang Hospital, Seongnam
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju
  - Yonsei University-Wonju Severance Christian Hospital, Wŏnju
- Spain (11):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario de La Ribera, Alzira
  - Hospital Universitario Reina Sofia, Córdoba
  - Complejo Hospitalario Ruber Juan Bravo, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital General de Segovia, Segovia
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - Vithas Hospital Sevilla, Seville
- Turkey (Türkiye) (8):
  - Ankara Universitesi Tip Fakultesi Hastanesi, Ankara
  - Adnan Menderes University Medical Faculty, Aydin
  - Dicle Üniversitesi, Diyarbakır
  - Erciyes University Medical Faculty, Kayseri
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi, Malatya
  - Mersin University, Mersin
  - Pamukkale University Medical Faculty, Fahri Goksin Oncology Centre, Pamukkale
  - Baskent University Dr. Turgut Noyan Research and Training Center, Yüreğir

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Daily Oral Orforglipron (LY3502970) Compared With Insulin Glargine in Participants With Type 2 Diabetes and Obesity or Overweight at Increased Cardiovascular Risk (ACHIEVE-4) — https://trials.lilly.com/en-US/trial/397395